CLINICAL TRIAL: NCT05706051
Title: Modification de la Posture et Appareillage Auditif Dans la Presbyacousie
Brief Title: Postural Modification and Hearing Aids in Presbycusis
Acronym: Post-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02002-41
Record Dates: First submitted 2022-12-05; First posted 2023-01-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Age-Related Hearing Loss; Postural; Defect; Hearing Aid
Keywords: Age-related hearing loss; presbycusis; posture; Hearing Aid
MeSH Terms: conditions — Presbycusis | interventions — Cytidine Diphosphate

STUDY DESIGN:
Intervention Model Description: Prospective study, with analysis of posturography parameters variation before and after hearing aid fitting in age-related hearing loss affected population aged 55 to 80 years old.
Masking Description: Ech individual is its proper control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- age-related hearing loss affected before hearing aid fitting (Other): patients aged 55 to 80 years old, undergoing posturography at diagnosis of ARHL and 3 months later before hearing aid fitting, within the role of control
  same patients udergoing posturography at hearing aid fitting and 3 months after.
  Interventions: Other: posturography

INTERVENTIONS:
Other: posturography — posturography will be performed when diagnosis of ARHL, in need of hearing aid fitting, is done and after information and written approval from patient. Posturography is performed later when hearing aid fitting and 3months after hearing aid use

SUMMARY:
Presbycusis could be associated to increased risk to fall. There is little about the impact on postural balance of hearing aids. In this study, the investigators describe the postural balance evolution before and after hearing aid fitting in presbycusis-affected adults (55-80years old) consulting Angers University Hospital ENT department and ENT Medical Doctor of Le Mans .

DETAILED DESCRIPTION:
After being informed about te study and consentment, patients meeting inclusion criteria consulting for presbycusis and in indication for hearing aids will be included to have posturometry (V0). Posturometry is performed 3 months later, before the first hearing aid installation (V1a) and after (V1b), as well as three months after hearing aid wearing (V2). Evolution of posturometry parameters without hearing aids between V0 and V1a serve as control and is compared to the evolution of posturometry parameters after hearing aid wearing between V1b and V2.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 80 years old
* ARHL within PTA superior to 30dBHL, and intelligibility threshold 30dB or worse defining hearing aid fitting indication in France

Non inclusion Criteria:

* hearing aid fitting refusal or contrindication
* vestibulare rehabilitation in past 3 months
* unusual physical activity the day of the posturography test
* incapacity to understand the instruction, or to stand up the time of posturography without help
* predictable incapacity to perform posturography in the time of the study

Exclusion criteria:

* acute affliction that could affect the posturography test
* daily physical activity modification due to medical advice or vestibular rehabilitation between two posturography

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Elliptic surface variation in posturography assessment before and after hearing aid fitting in presbycusis patients | 3 months
  analysis of variation of elliptic surface (cm2), eyes opened and closed, and subsequent romberg quotient (elliptic surface closed eyes/elliptic surface opened eyes) in the 3 months before hearing aid fitting and the 3 months after

SECONDARY OUTCOMES:
the effective wearing time of the device since its installation | 3 months
  average of time within hearing aid use per day (on the last 3 months)
the severity of the initial hearing loss | 3 months
  calculation of the average hearing loss measured by the average of the hearing thresholds without a hearing aid at 0.5, 1, 2 and 4 kHz
the notion of a balance disorder described by the patient | 3 months
  vertigo or feeling of instability

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Boucher, M.D., Ph.D., Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - UH Angers, Angers
  - Dr Lorin's otholaryngology practice, Le Mans

IPD SHARING:
Plan to Share IPD: Undecided
anonimized data within elliptic surface of posturography, PTA, and self reported dissiness